CLINICAL TRIAL: NCT04815590
Title: Pilot Study to Assess the Feasibility, Efficacy and Safety of Extended-release Injectable Buprenorphine for the Treatment of Opioid Use Disorder Among Individuals at High Risk of Overdose
Brief Title: Extended-release Injectable Buprenorphine for Individuals at High Risk of Overdose
Acronym: FASTER-BUP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BC Centre on Substance Use (Other)
Collaborators: Indivior Inc. (Industry)
Responsible Party: Principal Investigator, M. Eugenia Socias, Assistant Professor, Department of Medicine, UBC; Research Scientist, BCCSU, BC Centre on Substance Use
Other Study IDs: BCCSU-004
Record Dates: First submitted 2021-03-02; First posted 2021-03-25 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Opioid-Use Disorder; Opioid Overdose
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sublocade: The only group consists of participants with moderate to severe OUD who will be starting treatment with extended-release injectable buprenorphine as part of standard of care. While individual treatment regimens may vary, these will often consist of 2 once-monthly 300 mg subcutaneous injections followed by 4 once-monthly 100 mg subcutaneous injections. However, participants may receive once-monthly 300 mg subcutaneous injections in place of 100 mg subcutaneous injections for as many months as is deemed necessary by their prescribing physician.

SUMMARY:
This pilot study will evaluate the feasibility and clinical utility of extended-release injectable buprenorphine (XR-BUP) for the treatment of opioid use disorder (OUD) among individuals at high-risk for overdose (OD).

DETAILED DESCRIPTION:
FASTER-BUP is a 24-week observational pilot study evaluating the feasibility and clinical utility of XR-BUP (brand name: Sublocade) for the treatment of OUD among individuals at high-risk of OD. Forty participants with moderate to severe OUD starting treatment with XR-BUP as part of standard of care will be followed.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet ALL the following criteria to be eligible to participate for the study:

1. Be above 19 years of age;
2. Be diagnosed with moderate or severe OUD as evidenced by their approval for treatment with XR-BUP (Sublocade);
3. Be at high-risk for recurrent overdose, defined as having experienced a recent non-fatal overdose within the past 6 months (e.g., admission to the emergency department for an overdose OR self-reported OD that required Naloxone administration OR had an overdose where an ambulance arrived at the scene);
4. Have a new prescription for XR-BUP, but have not yet initiated treatment;
5. Be able and willing to follow study procedures;
6. Be able to provide adequate locator information (e.g., phone number and at least one emergency contact);
7. Be able and willing to provide written informed consent;
8. Be able to understand, communicate and speak with the research staff. Non-English speaking individuals will require a translator to be present during all study visits and during all study activities. The translator will be independent (e.g., not known to the participant to prevent the risk for coercion or misrepresentation).

Exclusion Criteria:

Participants will be excluded from the study if ANY of the following criteria are met:

1. Be on OAT other than buprenorphine/naloxone in the 7 days prior to screening;
2. Be on a stable buprenorphine/naloxone dose for more than 27 days prior to screening;
3. Use of an investigational drug in the 30 days prior to screening;
4. Incarcerated, pending legal action or other reasons that might prevent completion of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 40 eligible participants are planned to be enrolled into the study. Interested individuals must meet all of the inclusion criteria and none of the exclusion criteria to be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-10-17 (Estimated); Study Completion 2023-10-17 (Estimated)

PRIMARY OUTCOMES:
Number of XR-BUP injections received | 24 weeks
  The primary outcome for this study will be retention in treatment, defined as having received the six scheduled XR-BUP injections and completed the EOS/Early Termination visit.
Proportion of treatment-engaged visits per participant | 24 weeks
  Proportion of treatment-engaged visits per participant will be calculated as the number of received XR-BUP injections divided by the number of scheduled injections (i.e., six).

SECONDARY OUTCOMES:
Percentage of opioid free weeks | 24 weeks
  Suppression of illicit opioid use will be measured as the percentage of opioid-free weeks during the active treatment period (Visit 2 to Visit 8), using a combination of Urine Drug Test (UDT) results and self-reported illicit opioid use.
Safety monitoring | 24 weeks
  Descriptive statistics will be used for all safety analysis variables. No formal inferential tests will be performed on safety data.
  The incidence of all AEs will be summarized by body system, severity, seriousness, and relationship to the study drug using MedDRA. SAEs will be tabulated by patient.
  Descriptive statistics will be reported for injection site grading.

CONTACTS AND LOCATIONS:
Overall Officials: M. Eugenia Socias, MD, MSc., Principal Investigator — Assistant Professor, Department of Medicine, University of British Columbia
Locations (1):
- Rapid Access Addiction Clinic (RAAC), St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No